CLINICAL TRIAL: NCT05503316
Title: The Roll of Balance Confidence in Gait Rehabilitation in Persons With a Lesion of the Central Nervous System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2022-0324
Record Dates: First submitted 2022-08-04; First posted 2022-08-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Spinal Cord Injuries; Traumatic Brain Injury
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRAIL group (Experimental): Participants will receive 5 weeks of training on the GRAIL device, which is focused on training balance during walking.
  Therapy frequency: 2*30 minutes per week.
  Interventions: Other: Dynamic balance training
- Traditional gait rehabilitation (Active Comparator): Participant will receiver traditional gait rehabilitation which also includes training balance during walking.
  Therapy frequency in both groups is equal.
  Interventions: Other: Traditional gait rehabilitation

INTERVENTIONS:
Other: Dynamic balance training — Participants will receive dynamic balance training while walking on the GRAIL device.
  Arms: GRAIL group
Other: Traditional gait rehabilitation — Participants will receive traditional gait rehabilitation that also includes balance training while walking but not on the GRAIL device.
  Arms: Traditional gait rehabilitation

SUMMARY:
Persons with an injury of the central nervous system clearly experience motor impairments. Among the most commonly described consequences are gait abnormalities and impaired balance. Although these are undeniably linked, they are also influenced by other factors. A recent systematic review (Xie, 2022) reports impaired balance, the presence of depression or anxiety, and decreased function of the lower limbs as important risk factors for fear of falling in persons after a stroke. Also for people with a spinal cord injury, the fear of falling has a major impact on their level of participation and quality of life (Sing, 2021). Preventing falls and reducing fear of falling is an important part of neurological rehabilitation programs as it is known that fear of falling has a negative impact on the patient's activity level. This in turn will lead to an increased risk of falling and a negative effect on neurological recovery due to insufficiently practicing their balance while walking.

Since 2019 the rehabilitation center of UZ gent offers GRAIL training. This device aims to train walking balance and gait adaptability in a virtual environment. Patients who are admitted and/or undergoing ambulatory rehabilitation at UZ Gent are given the opportunity to complete a 5-week training schedule on the GRAIL. Before and after this training intervention period, the investigators evaluate the gait pattern of these patients. After the training period, the patients also complete a questionnaire about their experience while training on the GRAIL and often also indicate that they become more confident in their own balance when walking. That is why the researchers now also want to measure this.

Research questions:

1. Do people with high confidence in their balance when walking differ from those with low confidence in their balance when walking?
2. Does GRAIL training have a different effect on confidence in balance than traditional rehabilitation? To answer the 2nd research question, patients who follow the traditional rehabilitation (control group) also receive the same tests as the people who follow GRAIL training.

Randomization (prepared in advance via a computer program) determines who will follow the GRAIL training and who will follow the traditional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are admitted to the rehabilitation center of the Ghent University Hospital (in and outpatient) and suffered a stroke, spinal cord injury of traumatic brain injury
* Persons have to be able to walk for at least 6 minutes without the need of a person to help and with minimal help of a walking device. (level FAC 2 or higher)
* Participants who understand orders during the assessment and intervention.

Exclusion Criteria:

* Other neurological conditions (MS, Parkinson, ...)
* Orthopedic trauma or recent acute trauma that influence walking ability.
* Body weight exceeds 120 kg.
* Severe dizziness that makes it impossible to practice in standing position.
* Cardiac or pulmonary problems that require monitoring during exercising.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Gait speed (m/s) | Before the intervention
  Difference in gait speed between persons with high balance confidence and low balance confidence measured during walking on the treadmill.
Step length (m) | Before intervention
  Step length (m)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Step width (m) | Before intervention
  Step width (m)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Cadence (steps per minute) | Before intervention
  Cadence (steps per minute)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Cadence (steps per minute) | Within one week after the intervention
  Cadence (steps per minute)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Time in swing and stance phase (s) | Before intervention
  Time in swing and stance phase (s)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Time in swing and stance phase (s) | Within one week after the intervention
  Time in swing and stance phase (s)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Step width (m) | Within one week after the intervention
  step width (m)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
Step length (m) | Within one week after the intervention
  Step length (m)
  * Difference in spatiotemporal parameters between persons with high balance confidence and persons with low balance confidence (measured before intervention).
  * Difference in spatiotemporal parameters during normal walking and during a balance task during walking (measured before and after intervention period)
  * Difference in spatiotemporal parameters during normal walking before and after intervention.
10 meter walk test | Before intervention
  Difference in gait speed between persons with high balance confidence and low balance confidence measured during walking overground.
  Change in overground walking speed before and after intervention.
10 meter walk test | Within one week after the intervention
  Difference in gait speed between persons with high balance confidence and low balance confidence measured during walking overground.
  Change in overground walking speed before and after intervention.
Margins of stability | Before intervention
  Dynamic balance during walking measured during normal walking and during the balance task.
Margins of stability | Within one week after the intervention
  Dynamic balance during walking measured during normal walking and during the balance task.
Activity-specific Balance Confidence (ABC) scale | Before intervention
  Balance confidence scored by the participant (questionnaire) per item (16 items) geeft participant weer hoeveel vertrouwen hij heeft in dit item (0-100%) Hogere score is meer vertrouwen.
Activity-specific Balance Confidence (ABC) scale | Within one week after the intervention
  Balance confidence scored by the participant (questionnaire) per item (16 items) geeft participant weer hoeveel vertrouwen hij heeft in dit item (0-100%) Hogere score is meer vertrouwen.
Visual analogue scale score to assess task specific confidence | Before intervention
  Participants are asked to score the level of confidence that they have that they can complete the balance task (score 0-10).
  Higher score is more confidence.
Visual analogue scale score to assess task specific restraints | Before intervention
  Participants are asked to score the level of restraint that they have to complete the balance task due to fear of falling (score 0-10).
  Higher score is more restraint.
Visual analogue scale score to assess task specific confidence | Within one week after the intervention
  Participants are asked to score the level of confidence that they have that they can complete the balance task (score 0-10).
  Higher score is more confidence.Participants are asked to score the level of restraint that they have to complete the balance task due to fear of falling (score 0-10).
Visual analogue scale score to assess task specific restraints | Within one week after the intervention
  Participants are asked to score the level of restraint that they have to complete the balance task due to fear of falling (score 0-10).
  Higher score is more restraint.

SECONDARY OUTCOMES:
Quality of life using the SF36_C questionnaire | Before intervention
  Questionnaire to assess the quality of life (SF36_C)
  * Do persons with high balance confidence have better quality of life?
  * Does the quality of life change after the intervention?
Quality of life using the SF36_C questionnaire | Within one week after the intervention
  Questionnaire to assess the quality of life (SF36_C)
  * Do persons with high balance confidence have better quality of life?
  * Does the quality of life change after the intervention?
Anxiety and depression | Before intervention
  Hospital anxiety and depression scale (HADS)
  * Do persons with high balance confidence have less anxiety and depression?
  * Does the anxiety and depression change after the intervention?
Anxiety and depression | Within one week after the intervention
  Hospital anxiety and depression scale (HADS)
  * Do persons with high balance confidence have less anxiety and depression?
  * Does the anxiety and depression change after the intervention?
Gait quality | Within one week after the intervention
  Joint angles of lower limbs and trunk (degree) Do persons with high balance confidence walk different than persons with low balance confidence.
Scoring on a visual analogue scale to assess fear of falling | Before intervention
  Visual analogue scale (0-10) to indicate fear of falling during walking overground in the rehabilitation center and during walking on the treadmill.
  Higher score is more fear to fall.

CONTACTS AND LOCATIONS:
Overall Officials: Anke Van Bladel, PhD, Principal Investigator — Ghent University Hopsital / Ghent University
Locations (1):
- Ghent University Hospital, Ghent, Belgium